CLINICAL TRIAL: NCT04361630
Title: Recombinant Human Fibroblast Growth Factor-2 (rhFGF-2) In Absorbable Collagen Membrane With Coronally Advanced Flap In Class I And II Gingival Recession Defects -A Randomized Control Trial
Brief Title: Recombinant Human Fibroblast Growth Factor-2 (rhFGF-2) In Gingival Recession Defects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: SVS Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr R Viswa Chandra, Primary Investigator, SVS Institute of Dental Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SVSIDS/PERIO/3/2018
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Periodontitis
Keywords: Gingival Recession; Fibroblast Growth Factor 2; Periodontal Atrophy
MeSH Terms: conditions — Periodontitis; Gingival Recession; Periodontal Atrophy | interventions — Fibroblast Growth Factor 2

STUDY DESIGN:
Intervention Model Description: This study was a single-arm trial to obtain preliminary data on the efficacy of collagen membranes impregnated with recombinant human fibroblast growth factor (rhFGF-2) in the treatment of Miller's class I and class II gingival recessions.
Masking Description: Single Blinded trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main treatment group (Experimental): Collagen membranes incorporating 10ng/ml human recombinant basic fibroblast growth factor (FGF-2/bFGF) will be placed in the sites.
  Interventions: Drug: FGF 2

INTERVENTIONS:
Drug: FGF 2 — Following a standard surgical protocol, rhFGF-2 impregnated membranes will be placed in sites with gingival recession.
  Other Names: FGF+Collagen

SUMMARY:
This study was a single-arm trial to obtain preliminary data on the efficacy of collagen membranes impregnated with recombinant human fibroblast growth factor (rhFGF-2) in the treatment of Miller's class I and class II gingival recessions.

DETAILED DESCRIPTION:
Soft tissues can be regenerated to cover root exposure and a thin biotype can be converted into a thick biotype by using recombinant human growth factor technology. A recent review stated that growth factors could enhance soft tissue regeneration which includes restoration of mucogingival architecture and regeneration of periodontal hard and soft tissues including bone, cementum and periodontal ligament fibers. Fibroblast growth factor-2 (FGF-2), a heparin-binding cytokine with strong angiogenic activity stimulates the proliferation of undifferentiated mesenchymal cells. These functions can be applied in mucogingival surgery as FGF-2 promotes bone and cementum formation and exhibits an increased potential to promote periodontal regeneration in recession defects.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy subjects between 20-55 years presenting with Miller's class I or class II gingival recession[

Exclusion Criteria:

* 1. Recessions associated with root demineralization/caries, deep cervical abrasion or pulpal pathology, 2. Patients with history of systemic conditions affecting periodontium and, 3. Smokers.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Width of keratinized gingiva (wKG) | 5 months
  To assess the wKG, the mucogingival junction was identified visually as the border between the movable (alveolar mucosa) and immovable tissue (gingiva). The distance from the gingival margin to the mucogingival junction was considered as the Wkg.

CONTACTS AND LOCATIONS:
Locations (1):
- SVS Institute of Dental Sciences, Mahabubnagar, Hyderabad, Andhra Pradesh, India

IPD SHARING:
Plan to Share IPD: No
No current plans to share data with other researchers.